CLINICAL TRIAL: NCT05080959
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Dose Escalation and Optional Dose Expansion Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of CPL-01 in Postoperative Pain After Open Inguinal Herniorrhaphy
Brief Title: A Phase 2, Randomized, Double-Blind, Dose Escalation Study in Postoperative Pain Open Inguinal Herniorrhaphy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cali Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPL-01-201
Record Dates: First submitted 2021-08-14; First posted 2021-10-18 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2021-10

CONDITIONS: Inguinal Herniorrhaphy
MeSH Terms: interventions — Ropivacaine; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CPL-01 (Experimental): CPL-01 200mg, 400mg, 600mg
  Interventions: Drug: CPL-01
- Naropin (Experimental): 150mg
  Interventions: Drug: Naropin 150 MG Per 20 ML Injection
- Placebo (Experimental): 30mL normal saline (0.9%)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CPL-01 — Subjects will receive a single dose
  Other Names: Infiltration of study drug
  Arms: CPL-01
Drug: Naropin 150 MG Per 20 ML Injection — Subjects will receive a single dose
  Other Names: Infiltration of study drug
  Arms: Naropin
Drug: Placebo — Subjects will receive a single dose
  Other Names: Infiltration of study drug
  Arms: Placebo

SUMMARY:
This is a Phase 2b, randomized, double blind, placebo and active controlled study with an Ascending Dose Stage and an optional Dose Expansion Stage in subjects undergoing open inguinal herniorrhaphy with mesh.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo- and Active-Controlled, Dose Escalation and Optional Dose Expansion Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of CPL-01 in the Management of Postoperative Pain After Open Inguinal Herniorrhaphy.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to sign the informed consent form (ICF) prior to study participation.
* In the medical judgment of the Investigator, be a reasonably healthy adult 18 - 75 years of age, inclusive, and American Society of Anesthesiology (ASA) physical Class 1 or 2 at the time of randomization
* Plan to undergo an elective open inguinal herniorrhaphy with mesh under general anesthesia without collateral procedures or additional surgeries. Endotracheal intubation is not required.
* Have a body mass index ≤ 39 kg/m2.
* In the judgment of the Investigator, be willing and able to complete study procedures and pain scales and to communicate meaningfully with study personnel and return for outpatient follow-up visits as required.

Exclusion Criteria:

* Has previously undergone herniorrhaphy with the exception of a pediatric herniorrhaphy prior to 2 years of age.
* Has undergone 3 or more surgeries within 12 months prior to signing the ICF, other than for diagnostic procedures (e.g., colonoscopy).
* Has a history or clinical manifestation of significant medical, neuropsychiatric, or other condition including a clinically significant existing arrhythmia, bundle branch block or abnormal electrocardiogram (ECG), myocardial infarction or coronary arterial bypass graft surgery within the prior 12 months, significant abnormal clinical laboratory test value, or known bleeding abnormality that could preclude or impair study participation or interfere with study assessments.
* Has history or evidence of impaired liver function (e.g., ALT > 3 × upper limit of normal [ULN] or total bilirubin > 2 × ULN), active hepatic disease, or cirrhosis.
* Has history or evidence of impaired renal function (e.g., creatinine > 1.5 × ULN).
* Has a history of malignancy in the past year, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized in situ carcinoma of the cervix.
* Has or has had active COVID-19 infection within 3 months prior to surgery.
* Has a history of, or positive test results for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus antibody at Screening.
* Within 7 days prior to the scheduled surgery, be taking any central nervous system ( CNS) active agent as an analgesic adjunct medication, such as anticonvulsants, gabapentinoids, antidepressants (such as serotonin and norepinephrine reuptake inhibitors [SNRIs], selective serotonin reuptake inhibitors [SSRIs], and tricyclic antidepressants), benzodiazepines, sedative-hypnotics, clonidine and other central alpha-2 agents (e.g., tizanidine), ketamine, or muscle relaxants. These drugs are permitted if prescribed for non-pain indications and the dose has been stable for at least 30 days prior to surgery. The dose must remain stable throughout the study.
* Use of benzodiazepines and non-benzodiazepines (eszopiclone, ramelteon, zaleplon and zolpidem) is permitted to treat insomnia during the postoperative period.
* Within 7 days prior to the scheduled surgery and throughout the study, be taking antiarrhythmics except beta-blockers, digoxin, warfarin (see exception below), lithium, or aminoglycosides or other antibiotics for an infection (ophthalmic use or for treatment or prophylaxis of postoperative surgical site infections is permitted).
* Within 14 days prior to the scheduled surgery and throughout the inpatient period, be taking or using any cannabidiol-containing products, dietary supplements, or over-the- counter (OTC) preparations (e.g., chaparral, comfrey, germander, jin bu huan, kava, pennyroyal, skullcap, St. John's wort, or valerian).
* Within 28 days prior to the scheduled surgery, has received parenteral or oral corticosteroid treatment (steroid inhaler for allergy or asthma treatment, topical steroid for a non-clinically significant skin condition not involving the area of surgery or ophthalmic steroids are permissible).
* Is taking an antianginal, antihypertensive agent or diabetic regimen at a dose that has not been stable for at least 30 days or which is not expected to remain stable while participating in the study.
* In the opinion of the Investigator, within the past year has a history of illicit drug use or prescription medicine or alcohol abuse (regularly drinks > 4 units of alcohol per day, where 1 unit = 8 ounces beer, 3 ounces of wine, or 1 ounce of spirits).
* Has a positive alcohol breath/saliva test result indicative of alcohol use, or a positive urine drug screen result indicative of illicit drug use (unless results can be explained by a current prescription or acceptable OTC medication at Screening as determined by the Investigator) at Screening and/or prior to surgery.
* Has previously participated in a clinical study with CPL-01.
* Has participated in another clinical trial or used an investigational product within 30 d days or 5 half-lives, whichever is longer, prior to the planned surgery or is scheduled to receive any other investigational product while participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
AUC of the NRS-A for pain (Primary Endpoint) | 0 - 72 hours
  Summary (area under the curve) through 72 hours of the Numeric rating scale with activity score for pain, where 0 is no pain and 10 is worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Erol Onel, MD, Study Chair — Cali Biosciences
Locations (5):
- United States (5):
  - Shoals Medical Trials, Inc, Sheffield, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - First Surgical Hospital, Bellaire, Texas
  - Jean Brown Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No